CLINICAL TRIAL: NCT01839396
Title: Implantable Neurostimulator for the Treatment of Parkinson's Disease
Brief Title: Deep Brain Stimulation (DBS) for the Treatment of Parkinson's Disease
Acronym: INTREPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G120075; CDM00049710/90876693 (Other: BSC protocol number)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Parkinson's Disease
Keywords: Intrepid, Vercise, PD, DBS, Boston Scientific
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medium continuous dose of stimulation (Active Comparator): Subjects in this arm will receive stimulation settings at a medium continuous dose of Deep Brain stimulation that may have been effective in previous DBS patients.
  Interventions: Device: Deep Brain Stimulation
- Low intermittent dose of stimulation (Sham Comparator): Subjects in this arm will receive stimulation settings at a lower intermittent dose of Deep Brain stimulation which is less likely to be effective.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — The Vercise™ DBS system will be implanted in subjects in both study arms. Stimulation parameters will vary depending on the study arm assignment. All subjects will receive therapeutic settings at the end of the blinded period.
  Other Names: Vercise™ Deep Brain Stimulation (DBS) system.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Boston Scientific's Vercise Deep Brain Stimulation (DBS) system in the treatment of patients with with advanced, levodopa-responsive bilateral Parkinson's disease (PD) which is not adequately controlled with medication.

DETAILED DESCRIPTION:
The study is multi-center, prospective, double-blind, randomized (3:1) controlled trial.

GUIDE XT may be used for planning of programming as needed.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of bilateral idiopathic PD (H&Y ≥ 2) with a duration of PD ≥ 5 years.
* Persistent disabling Parkinson's disease symptoms or drug side effects (e.g., dyskinesias, motor fluctuations, or disabling "off" periods) despite optimal medical therapy.
* Able to understand the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.

Key Exclusion Criteria:

* Any intracranial abnormality or medical condition that would contraindicate DBS surgery.
* Have any significant psychiatric condition likely to compromise the subject's ability to comply with requirements of the study protocol
* Any other active implanted devices including neurostimulators and /or drug delivery pumps
* Any previous thalamotomy, pallidotomy or subjects who have undergone a DBS procedure.
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
* A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Vitek, MD, PhD, Principal Investigator — University of Minnesota, Neurology Department; Philip Starr, MD, PhD, Principal Investigator — Universiry of California, San Francisco, Surgical Movement Disorders Clinic
Locations (22):
- United States (22):
  - Muhammad Ali Parkinson Research Center and Movement Disorders Clinic, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente, Sacramento, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Carepoint, PC d/b/a Blue Sky Neurology, Englewood, Colorado
  - University of Florida Shands Hospital, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - University of Miami, School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Albany Medical Center, Albany, New York
  - NYU Medical Center, New York, New York
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Vitek JL, Jain R, Chen L, Troster AI, Schrock LE, House PA, Giroux ML, Hebb AO, Farris SM, Whiting DM, Leichliter TA, Ostrem JL, San Luciano M, Galifianakis N, Verhagen Metman L, Sani S, Karl JA, Siddiqui MS, Tatter SB, Ul Haq I, Machado AG, Gostkowski M, Tagliati M, Mamelak AN, Okun MS, Foote KD, Moguel-Cobos G, Ponce FA, Pahwa R, Nazzaro JM, Buetefisch CM, Gross RE, Luca CC, Jagid JR, Revuelta GJ, Takacs I, Pourfar MH, Mogilner AY, Duker AP, Mandybur GT, Rosenow JM, Cooper SE, Park MC, Khandhar SM, Sedrak M, Phibbs FT, Pilitsis JG, Uitti RJ, Starr PA. Subthalamic nucleus deep brain stimulation with a multiple independent constant current-controlled device in Parkinson's disease (INTREPID): a multicentre, double-blind, randomised, sham-controlled study. Lancet Neurol. 2020 Jun;19(6):491-501. doi: 10.1016/S1474-4422(20)30108-3. Epub 2020 May 26. PMID 32470421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were considered enrolled once informed consent was completed. Only those who met all eligibility criteria went on to receive implant and randomization for study endpoints
Pre-assignment Details: Subjects were considered enrolled once informed consent was completed. Only those who met all eligibility criteria went on to receive implant and randomization for study endpoints
Groups:
- Medium Continuous Dose of Stimulation: Subjects in this arm received a medium continuous dose of Deep Brain stimulation that may have been effective in previous DBS patients.
  Deep Brain Stimulation: The Vercise™ DBS system was implanted in subjects in both study arms. Stimulation parameters varied depending on the study arm assignment. All subjects received therapeutic settings at the end of the blinded period.
- Low Intermittent Dose of Stimulation: Subjects in this arm received a lower intermittent dose of Deep Brain stimulation which was less likely to be effective.
  Deep Brain Stimulation: The Vercise™ DBS system was implanted in subjects in both study arms. Stimulation parameters varied depending on the study arm assignment. All subjects received therapeutic settings at the end of the blinded period.
Period: Overall Study
Arm/Group | Medium Continuous Dose of Stimulation | Low Intermittent Dose of Stimulation
Started | 121 | 39
Completed | 121 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medium Continuous Dose of Stimulation | Low Intermittent Dose of Stimulation | Total
Number analyzed (Participants) | 121 | 39 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age is reported at time of enrollment Population: Information for each group and overall population is provided.
  years
    Age | 60.7 (7.9) | 57.5 (7.66) | 59.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 13 | 44
  Male | 90 | 26 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change in ON Time as Measured by Parkinson's Disease Diary
Description: Difference in the mean change from baseline to 12 weeks post-randomization between the active and control groups in the ON time as measured by Parkinson's diary. Positive indicates improvement
Time Frame: From baseline to 12 weeks post-randomization
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Medium Continuous Dose of Stimulation: Subjects in this arm received a medium continuous dose of Deep Brain stimulation that may have been effective in previous DBS patients.
  Deep Brain Stimulation: The Vercise™ DBS system was implanted in subjects in both study arms. Stimulation parameters were varied depending on the study arm assignment. All subjects received therapeutic settings at the end of the blinded period.
- Low Intermittent Dose of Stimulation: Subjects in this arm received a lower intermittent dose of Deep Brain stimulation which was less likely to be effective.
  Deep Brain Stimulation: The Vercise™ DBS system was implanted in subjects in both study arms. Stimulation parameters were varied depending on the study arm assignment. All subjects received therapeutic settings at the end of the blinded period.
Arm/Group | Medium Continuous Dose of Stimulation | Low Intermittent Dose of Stimulation
Number analyzed (Participants) | 118 | 38
hours | 3.74 (4.79) | 0.72 (3.56)

2. Secondary Outcome: Secondary Endpoints
Description: Change in Unified Parkinson's Disease Rating Scale (UDPRS) Part III (stim on/meds off) from baseline to 12 weeks post randomization.
  Range of UPDRS III is 0 - 108 with greater scores indicating worse disease state.
Time Frame: From baseline to 12 weeks post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medium Continuous Dose of Stimulation | Low Intermittent Dose of Stimulation
Number analyzed (Participants) | 115 | 37
units on a scale | 12.02 (11.4) | 1.19 (8.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 12 weeks and up to Dec 2016.
Description: Serious Adverse Events related to hardware, stimulation or procedure are reported
Arm/Group | Medium Continuous Dose of Stimulation | Low Intermittent Dose of Stimulation
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/39
Serious Adverse Events (participants affected / at risk) | 14/121 | 4/39
Other Adverse Events (participants affected / at risk) | 35/121 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medium Continuous Dose of Stimulation (N=121) | Low Intermittent Dose of Stimulation (N=39)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Confusional postoperative (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Convulsion (Psychiatric disorders) | 1 (1) | 1 (1)
Device related Infection (Infections and infestations) | 3 (3) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Implant Site Edema (General disorders) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Staphylococcal Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Heamorhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medium Continuous Dose of Stimulation (N=121) | Low Intermittent Dose of Stimulation (N=39)
Balance Disorder (Nervous system disorders) | 7 (7) | 0 (0)
Dyskinesia (Nervous system disorders) | 21 (23) | 1 (1)
Implant Site Edema (General disorders) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement that restricts the PIs until official study manuscript is published.